CLINICAL TRIAL: NCT05371561
Title: Influence of Different Personal Protective Equipment on Children's Fear in Dental Office: A Randomized Controlled Trial
Brief Title: Effect of PPE on Children's Fear in Dental Office
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maha Moussa Azab, Lecturer, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Fayoum U
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Infections; COVID-19 Virus Infection
Keywords: PPE; Dentist attire; Child behavior; dental fear
MeSH Terms: conditions — COVID-19; Infections; Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants, legal guardians, and the dentist who carried out the examination were not blinded as it was inapplicable. The accessor and statistician were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Goggles + surgical mask (Active Comparator): Dentist wearing Goggles + surgical mask will examin the patient
  Interventions: Device: reusable respirators
- Face shield+ surgical mask (Active Comparator): Dentist wearing Face shield+ surgical mask will examin the patient
  Interventions: Device: reusable respirators
- Half face reusable respirator+ Filter (Experimental): Dentist wearing Half face reusable respirator+ Filter will examin the patient
  Interventions: Device: reusable respirators
- Full face reusable respirator+ Filter (Experimental): Dentist wearing Full face reusable respirator+ Filter will examin the patient
  Interventions: Device: reusable respirators

INTERVENTIONS:
Device: reusable respirators — Dentist wearing reusable respirator will examin the patient

SUMMARY:
the aim of the current study is to compare the effect of conventional facial PPE as 1)goggles + surgical masks, and 2)face shields + surgical masks versus 3)half-face and 4)full-face reusable respirators; on preoperative child's fear in the dental office.

DETAILED DESCRIPTION:
Each patient meeting the inclusion criteria and assigned to a specific study group will enter the clinic for dental examination. The examining dentist, wearing the selected PPE will communicate with patient and parent, taking personal, previous and current history, and carrying out simple examination not involving the use of sharp instruments, provoking pain or investigations as radiographs. The process should take from three to five minutes. Then, the child will be escorted to another room to meet a blinded accessor, where he assesses the child's anxiety using the Arabic version of children's fear survey schedule-dental subscale CFSS-DS.

ELIGIBILITY:
Inclusion Criteria:

* Six to ten-year-old patients

Exclusion Criteria:

* emergency patients
* patients who have systemic, mental or psychological conditions as indicated by their medical history,

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Arabic version of children's fear survey schedule-dental subscale (CFSS-DS) | just after examination
  Children's fear survey schedule-dental subscale CFSS-DS is a tool to measure children's anxiety in dental settings. The CFSS-DS consists of 15 items, revolving around dental setting and procedures, child will answer each item by choosing a rate from a 5-point Likert scale that ranges from 1 ('not afraid at all') to 5 ('very afraid'), the total score should range from 15 to 75

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azab MM. Influence of different personal protective equipment on children's anxiety in dental office: a randomized controlled trial. BMC Oral Health. 2022 Sep 22;22(1):421. doi: 10.1186/s12903-022-02442-5. PMID 36138354